CLINICAL TRIAL: NCT00223431
Title: Clinical Performance of Three-Unit Fixed Partial Dentures (FPDs) Made From a Hot-Pressed Ceramic (Five-Year Study)
Brief Title: Clinical Performance of 3-Unit FPDs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114-1998
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Partial Edentulism

INTERVENTIONS:
Device: all-ceramic fixed partial denture

SUMMARY:
Objectives: The purpose of this research was to determine the clinical success rate of a lithia-disilicate-based core ceramic (Ivoclar, Vivadent Corp.) for use in posterior fixed partial dentures (FPDs) as a function of bite force, cement type, connector height, and connector width.

Methods: Thirty ceramic FPD core frameworks were prepared using a hot-pressing technique and a lithia-disilicate-based core ceramic. The maximum clenching force was measured for each patient prior to tooth preparation. Connector heights and widths were measured for each FPD. Patients were recalled yearly after cementation for two years and evaluated using eleven clinical criteria. All FPDs were examined by two independent clinicians and rankings for each criterion were made from 1 to 4 with 4 = excellent and 1 = unacceptable.

The aims of this research were:

1. To test the hypotheses that three-unit fixed partial dentures (FPDs) of a high-strength core ceramic will exhibit good-to-excellent clinical performance (based on 11 evaluative criteria) and that they will adequately resist fracture in posterior situations (excluding third molars) if fabricated with the minimal connector size (4 mm x 4 mm).
2. To test the hypothesis that a reinforced glass ionomer cement (ProTec CEM, Ivoclar, Vivadent), when used to cement core ceramic crowns in posterior FPDs, will be associated with significantly less marginal quality, but similar fracture resistance of the ceramic crowns compared with the marginal quality associated with a dual cure resin cement (Variolink® II, Ivoclar Vivadent AG, Schaan, Liechtenstein).
3. To test the hypothesis that there is no significant difference in tooth sensitivity associated with FPDs cemented with the glass ionomer cement and dual-cure resin cement.

DETAILED DESCRIPTION:
All patient recruitment and treatment were performed at the University of Florida College of Dentistry, Graduate Prosthodontic Clinic by Prosthodontic faculty. Patients were initially screened to exclude individuals with medical contraindications to dental treatment, parafunctional habits, and inability to ensure residence in the area for the next five years. Inclusion criteria were a missing posterior tooth in a quadrant (first premolars through second molars) that could be restored with a 3-unit FPD, periodontal pockets of less than 4 mm for each abutment with no periodontal disease, vital abutment teeth, and a crown root ratio of at least 1:1. A patient can have multiple FPDs placed as long as the above-mentioned criteria were met. Baseline data were obtained for each selected subject to include the following:

1. General medical history and physical examination
2. Primary casts made with irreversible hydrocolloid impression material
3. Bite force measurement in Newtons made with a gnathodynamometer
4. Pocket depths of abutment teeth
5. Periapical radiographs of abutment teeth. The maximum occlusal force exerted by each subject was measured prior to commencing treatment using a bite force gauge that has been reported previously by Gibbs et al.12 The purpose of these measurements was to analyze the influence of occlusal force on the survival of the FPDs. A total of 30 FPDs were fabricated for 21 patients with the core ceramic and all patients were recalled each year for two years. Three clinicians performed treatment and one technician using an in-house laboratory accomplished all labwork. Out of the 21 patients, 18 were female and 3 were male with ages ranging from 30 to 62 years of age. The 3-unit FPDs were located in the posterior area with canines serving as the most anterior abutment and second molars as the most posterior abutment. All FPDs were opposed by natural dentition. The dimensions for tooth reduction included at least 1 mm of axial reduction; 2 mm of occlusal reduction and incorporation of a shoulder or a deep chamfer margin design with rounded line angles. Final impressions were made using a dual impression technique with high and low viscosity polyvinylsiloxane in a stock tray. Provisional resin FPDs were made and cemented with temporary cement. FPDs were processed by hot-pressing the core ceramic (Ivoclar Vivadent AG, Schaan, Liechtenstein) and applying stain and glaze as necessary. The heat-pressed ceramic system uses the lost wax technique whereby the FPD is waxed to its proper shape and contour and then invested in a special flask with a special type of investment material. The desired shade of a precerammed ceramic cylinder is plasticized at 1100oC and pressed under vacuum and pressure into the mold of the investment.13 The ceramic FPDs were inspected to ensure that the incisogingival height and curvature of the gingival embrasure of the connectors were adequate to resist fracture when subjected to normal biting forces. The minimal dimensions recommended for premolar FPDs, 4 mm x 4 mm, and for molar FPDs, 4 mm x 5 mm, were applied for each FPD when esthetics and gingival contour permitted. Connector heights and widths were measured for each FPD using a boley gauge. FPDs were cemented using either a resin-reinforced glass ionomer cement (Protec CEM, Vivadent) or a dual-cure resin cement (Variolink II, Vivadent) using a random number table. Fourteen (14) FPDs were cemented with the resin-reinforced glass ionomer and 13 with the dual cure resin. Patients were recalled after cementation annually for two years and evaluated for the following clinical criteria: (1) tissue health; (2) secondary caries; (3) occlusion; (4) proximal contact; (5) marginal integrity; (6) absence of sensitivity to percussion, heat, cold, and air; (7) color match; (8) surface texture; (9) absence of wear of opposing teeth; (10) anatomic contour; and (11) no cracks/chips or fracture. This evaluative system was derived from the California Dental Association quality assessment evaluation system.14 FPDs were examined by two independent clinicians who did not prepare the teeth or cement the prosthesis, and rankings of each criterion were made from 1 to 4 with 4 = excellent, 3 = good, 2 = unacceptable (needs repair or replacement in the near future), and 1 = unacceptable (needs immediate replacement). All clinicians/evaluators were subjected to several calibration exercises that consisted of table top analysis of marginal openings as well as slide evaluations of different clinical situations.

Data were analyzed by logistic regression analysis of the variables with α = 0.05. The consistency of the examiners' scores was evaluated for consistency using a test for the standard deviation of inter-examination.

ELIGIBILITY:
Inclusion Criteria:

* missing posterior tooth in a quadrant (first premolars through second molars) that could be restored with a 3-unit FPD
* periodontal pockets of less than 4 mm for each abutment with no periodontal disease
* vital abutment teeth
* crown root ratio of at least 1:1.

Exclusion Criteria:

* individuals with medical contraindications to dental treatment
* parafunctional habits
* inability to ensure residence in the area for the next five years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1998-02; Study Completion 2004-05

PRIMARY OUTCOMES:
clinical performance
improved esthetics
improved occlusal function of a lithia disilicate based core ceramic. Performance was measured yearly for 4 years.

SECONDARY OUTCOMES:
wear of opposing enamel

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Anusavice, PhD, DMD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Dentistry, Gainesville, Florida, United States

REFERENCES:
- [Result] Esquivel-Upshaw JF, Anusavice KJ, Young H, Jones J, Gibbs C. Clinical performance of a lithia disilicate-based core ceramic for three-unit posterior FPDs. Int J Prosthodont. 2004 Jul-Aug;17(4):469-75. PMID 15382785
- [Result] Gibbs CH, Anusavice KJ, Young HM, Jones JS, Esquivel-Upshaw JF. Maximum clenching force of patients with moderate loss of posterior tooth support: a pilot study. J Prosthet Dent. 2002 Nov;88(5):498-502. doi: 10.1067/mpr.2002.129062. PMID 12473999